CLINICAL TRIAL: NCT05729048
Title: Starling Continuous Renal Replacement Therapy (CRRT) Observational Study
Brief Title: Starling/CRRT Observational Study
Status: Withdrawn | Type: Observational
Why Stopped: Study Sponsor decided not to move forward with this project.
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU578332
Record Dates: First submitted 2022-11-29; First posted 2023-02-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hemodynamic Monitoring
Keywords: Cardiac Index (CI); Stroke Volume (SV); Stroke Volume Index (SVI); Stroke Volume Variation (SVV); Heart Rate (HR); Ventricular Ejection Time (VET); Total Peripheral Resistance (TPR); Total Peripheral Resistance Index (TPRI); Cardiac Power (CP); Cardiac Power Index (CPI); Blood Oxygenation (SPO2); Oxygen Delivery Index (DO2I); Electrical impedance of the chest cavity (Z0); Thoracic Fluid Content (TFC); Thoracic Fluid Content change from preset time period (TFCd); Thoracic Fluid Content from baseline (TFCd0); Changes in SV, CO and other hemodynamic parameters which are derived by Bioreactance® as a result of posture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemodynamic Monitoring: Over the course of a patient's hospitalization, data will be collected on patients from the initiation to completion of hemodynamic monitoring with the Starling monitor during CRRT treatment.
  Interventions: Device: Starling

INTERVENTIONS:
Device: Starling — Starling is a portable, non-invasive, cardiac output detector system. The Starling monitor measures the cardiac output by employing electrical bioreactance. Bioreactance is a measure of the electrical characteristics of a volume of tissue and fluid. In the case of cardiac output measurements, the relevant tissue includes the heart and the immediate surrounding volume of the thorax. The relevant fluid is blood.
  The Starling electrode is a double electrode sensor. Within each sensor, one electrode is used to transmit a high frequency sine wave into the body, while the resulting voltage is measured at the adjacent electrode.
  This information is used to determine cardiac output. The Starling monitor also measures and displays associated hemodynamic parameters based on calculations of measurements already incorporated into the Starling monitor.

SUMMARY:
Hemodynamic optimization of critically ill patients is a goal for clinicians in order to afford the patient the best possible outcomes. Being able to precisely and rapidly determine patient fluid responsiveness provides the bedside physician and nursing staff the information needed to make critical decisions in regard to the patient's fluid status and management of additional fluids and medications.

As fluid management and cardiac output determination are linked to better decision-making and improved outcomes in ICU, the use of a dynamic assessment of fluid responsiveness becomes a key tool for patient management.

This study is designed to collect treatment and outcome data on patients that have undergone hemodynamic monitoring during CRRT therapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 to 95 years of age.
2. Patient has undergone hemodynamic monitoring with the Starling monitor during a CRRT treatment.
3. Hemodynamic monitoring was completed no earlier than 2018

Exclusion Criteria:

1. Patients did not have an arterial line in place during CRRT treatment
2. Patients on extracorporeal membrane oxygenation (ECMO) or left ventricular assist device (LVAD)
3. Patients with end-stage kidney disease on chronic dialysis
4. Hemodynamic monitoring with Starling did not occur during CRRT treatment
5. Data from Starling, CRRT machine, or arterial line cannot be retrieved

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is defined as all patients who meet the study eligibility criteria and have undergone monitoring with the Starling monitor during CRRT. All available data will be included in the analysis.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in stroke volume (SV) after CRRT initiation | Day 1 (during CRRT)
Change in cardiac output (CO) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in cardiac index (CI) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in stroke volume (SV) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in stroke volume index (SVI) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in Thoracic Fluid Content (TFC) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in heart rate (HR) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in systolic blood pressure (SBP) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in diastolic blood pressure (DBP) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in central venous pressure (CVP) after fluid removal | Day 1 (during CRRT)
  Cardiac physiology adjusted to net ultrafiltration intensities (ml/kg/h)
Change in mixed venous oxygen saturation (SVO2) after fluid removal | Day 1 (during CRRT)
  Perfusion parameter adjusted to net ultrafiltration intensities (ml/kg/h)
Change in lactate after fluid removal | Day 1 (during CRRT)
  Perfusion parameter adjusted to net ultrafiltration intensities (ml/kg/h)
Changes in systolic blood pressure (SBP) from beginning to end of CRRT | Day 1 (Begin CRRT) through Day 1 (End of CRRT)
Changes in diastolic blood pressure (DBP) from beginning to end of CRRT | Day 1 (Begin CRRT) through Day 1 (End of CRRT)
Changes in mean arterial pressure (MAP) from beginning to end of CRRT | Day 1 (Begin CRRT) through Day 1 (End of CRRT)

SECONDARY OUTCOMES:
Incidence of intradialytic hypotension (IDH) during CRRT | Day 1 (during CRRT)
Incidence of intradialytic hypotension (IDH) free time during CRRT | Day 1 (during CRRT)
Incidence of time to resolution in intradialytic hypotension (IDH) during CRRT | Day 1 (during CRRT)
Changes in intake and output (I/O) during CRRT | Day 1 (during CRRT)
  Fluid balance parameter
Changes in hourly/daily fluid balance during CRRT | Day 1 (during CRRT)
Changes in cumulative fluid balance during CRRT | Day 1 (during CRRT)
Changes in percent fluid overload during CRRT | Day 1 (during CRRT)
  Fluid balance parameter
Changes in ultrafiltration parameters and net ultrafiltration (UFnet) during CRRT | Day 1 (during CRRT)
Incidence of ultrafiltration failure during CRRT | Day 1 (during CRRT)
  Including prescribed/archived, time to fluid balance
Blood flow rate during CRRT | Day 1 (during CRRT)
CRRT dose/modality | Day 1 (during CRRT)
Estimate the contribution degree of certain patient conditions, clinical characteristics, fluid, and CRRT parameters in predicting the IDH risk during CRRT | Day 1 (during CRRT)
Identify sub-phenotypes of patients at risk of IDH during CRRT | Day 1 (during CRRT)

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Investigational Site, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy